CLINICAL TRIAL: NCT00291694
Title: A Double-blinded Phase II Study of the Expression of Ki-67/MIB-1 in Women With Hyperplasia of the Breast Randomized to Receive Daily Celecoxib 400 mg BID or Placebo
Brief Title: Protocol for Women at Increased Risk of Developing Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carol Fabian, MD (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9118
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Results first posted 2013-09-05 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: breast atypia; double-blind randomized clinical trial; RCT; celecoxib; COX-2 inhibitor; placebo; high risk for breast cancer; breast epithelial hyperplasia; ki-67; chemoprevention
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Oral Celecoxib 400 mg twice daily for 12 months
  Interventions: Drug: celecoxib
- 2 (Placebo Comparator): Matched blinded placebo twice daily for 12 months
  Interventions: Other: placebo

INTERVENTIONS:
Drug: celecoxib — Celecoxib 400 mg BID
  Other Names: Celebrex
  Arms: 1
Other: placebo — placebo
  Arms: 2

SUMMARY:
To assess the effects of twelve months of celecoxib administration by evaluating breast tissue needle aspirations, to determine if cell growth can be slowed.

DETAILED DESCRIPTION:
A blind randomized study of celecoxib in women at high risk of developing breast cancer. Subjects are to take twelve months of drug/placebo. At baseline and after twelve months subjects will have a random periareolar fine needle breast aspiration that will be assessed for epithelial cell growth and other markers of risk. Baseline and twelve month serum samples will also be assessed for hormones and growth factors which may be associated with breast cancer risk. Mammograms at baseline and twelve months will also be assessed for breast density changes.

ELIGIBILITY:
Inclusion Criteria:

* women who have a high risk of breast cancer
* older than 18 years

Exclusion Criteria:

* anticoagulants
* marked breast tenderness
* pregnant or within twelve months of breast feeding/childbirth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo for 12 months
- Celecoxib: Celecoxib for 12 months
Period: Overall Study
Arm/Group | Placebo | Celecoxib
Started | 24 | 48
Completed | 21 | 43
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Celecoxib: Celecoxib for six months
- Placebo: Placebo for six months
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Placebo | Total
Number analyzed (Participants) | 48 | 24 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 24 | 72
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (6.6) | 45.2 (8.5) | 47.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 24 | 72
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 48 | 24 | 72

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent of Breast Epithelial Cells Staining Positive for Ki-67
Description: Immunocytochemical staining of breast epithelial cells. Positive cells reflect proliferative activity.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: percentage of cells staining positive
Groups:
- Celecoxib: Randomized to receive celecoxib daily for 12 months
- Placebo: Randomized to receive placebo daily for 12 months
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 43 | 21
percentage of cells staining positive | -1.2 [-18 to 14.8] | -2.0 [-8.8 to 12.2]
Statistical Analysis 1: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.71, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Mammographic Breast Density
Description: The percent of mammographic breast area that is considered to be at increased density. Evaluated using the semi-automated computer program Cumulus.
Time Frame: Baseline and 12 months
Population: Subjects completing 12 months, with baseline and 12 month mammograms suitable for density analysis, such that a change in density over time can be computed
Measure: Median (Standard Error); unit: percentage of breast area at increased d
Groups:
- Celecoxib: Oral Celecoxib 400 mg twice daily for 12 months
  celecoxib: Celecoxib 400 mg BID
- Placebo: Matched blinded placebo twice daily for 12 months
  placebo: placebo
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 44 | 19
percentage of breast area at increased d | -1.3 (1.0) | 0.3 (1.9)
Statistical Analysis 1: Comparison: Celecoxib vs Placebo; Difference between groups, two-sided. Endpoint not specifically powered for effect; Test type: Superiority or Other; p = 0.053, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons

3. Secondary Outcome: Serum Estradiol Concentration
Description: Change in serum estradiol concentration
Time Frame: Baseline to 12 months
Measure: Median (Standard Error); unit: pg/ml
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 43 | 21
pg/ml | -6.6 (5.9) | -5.7 (11.7)
Statistical Analysis 1: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons

4. Secondary Outcome: Serum Sex Hormone Binding Globulin (SHBG) Concentration
Description: Change in serum concentration
Time Frame: Baseline to 12 months
Measure: Median (Standard Error); unit: nmol/L
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 43 | 21
nmol/L | -0.70 (1.61) | 3.05 (2.16)
Statistical Analysis 1: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.39, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons

5. Secondary Outcome: Molecular Ratio of Serum Concentration of IGF-1 to IGFBP3
Description: Change ion ratio.
Time Frame: baseline to 12 months
Measure: Median (Standard Error); unit: ratio
Arm/Group | Celecoxib | Placebo
Number analyzed (Participants) | 43 | 21
ratio | -0.012 (0.0039) | -0.011 (0.0071)
Statistical Analysis 1: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Placebo: Randomized to receive palcebo daily for 12 months
Arm/Group | Celecoxib | Placebo
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/21
Other Adverse Events (participants affected / at risk) | 43/43 | 21/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Celecoxib (N=43) | Placebo (N=21)
Allergic Reaction (Immune system disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 5 (5) | 0 (0)
Fever (General disorders) | 2 (2) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 6 (6)
Skin-other (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Hot Flashes (Reproductive system and breast disorders) | 5 (5) | 3/12 (3)
Reproductive-other (Reproductive system and breast disorders) | 13 (13) | 3 (3)
Constipation (Gastrointestinal disorders) | 11 (11) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 18 (18) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 14 (14) | 5 (5)
Flatulence (Gastrointestinal disorders) | 13 (13) | 8 (8)
Nausea (Gastrointestinal disorders) | 7 (7) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
GI-other (Gastrointestinal disorders) | 8 (8) | 3 (3)
Rectal bleeding (Gastrointestinal disorders) | 4 (4) | 1 (1)
Infection-other (Immune system disorders) | 24 (24) | 13 (13)
Insomnia (Nervous system disorders) | 1 (1) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 10 (10) | 3 (3)
headache (Nervous system disorders) | 19 (19) | 6 (6)
pain-other (Nervous system disorders) | 19 (19) | 7 (7)
Pulmnary-other (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Renal-other (Renal and urinary disorders) | 0 (0) | 3 (3)
Irregular menses (Reproductive system and breast disorders) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes